CLINICAL TRIAL: NCT02073708
Title: A Population-based Investigation of Asthma in the Telemark Region of Norway
Status: Active, not recruiting | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Oslo University Hospital (Other); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency); Göteborg University (Other)
Responsible Party: Principal Investigator, Anne Kristin M. Fell, MD, PhD, Sykehuset Telemark
Other Study IDs: 1665
Record Dates: First submitted 2014-02-20; First posted 2014-02-27 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Lung Diseases; Respiratory Symptoms; Inflammation
MeSH Terms: conditions — Lung Diseases, Obstructive; Signs and Symptoms, Respiratory; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, citrate plasma, EDTA-plasma, whole blood, gene sequencing (next generation gene sequencing)
Oversight: Data Monitoring Committee: No

SUMMARY:
Respiratory conditions impose an enormous burden on the individual and the society. According to the WHO World Health Report 2000, the top five respiratory diseases - including asthma and COPD - account for 17% of all deaths and 13% of all Disability-Adjusted Life Years (DALYs). Obstructive lung diseases are among the most common chronic diseases in working-aged populations affecting ~40 million individuals in Europe. The greatest economic burden of respiratory diseases on health services and lost production in the EU is due to COPD and asthma, at about €20 billion each for healthcare and €25 billion and €15 billion, respectively, for lost production.

For Norway, there are no estimates of asthma prevalence for the country as a whole, but 80/1000 women and 55/1000 men used asthma medication in 2013 according to the national prescription register. Estimated annual deaths in Norway due to COPD were 4070 in 2015, which is 30% higher than for lung cancer. Unfortunately, a substantial proportion of patients are still difficult to treat. This underlines the need for better primary prevention and more knowledge regarding causes and exacerbating factors.

Several risk factors for chronic respiratory diseases are identified, most important tobacco smoke, closely followed by air pollution and occupational exposure. However, according to recent reviews there is a lack of understanding regarding environmental risk factors and mechanisms of how these affect respiratory health, the importance of biological markers and comorbidity, and of socioeconomic risk factors. Moreover, there is a need for assessment of interactions between risk factors and between the individual and the environment.

Telemark has a high proportion of craft- and industrial workers providing exposure contrasts. Furthermore, the use of medication against respiratory diseases and the rate of sick leave are higher in Telemark than elsewhere in Norway. Moreover, the county has a high rate of disability. There are previous studies from other parts of Norway, which have estimated the occurrence of respiratory diseases and provided valuable knowledge regarding some risk factors. However, these studies use crude measures of self-reported exposure and do not provide sufficient information on how to target intervention and implement effective prevention. In contrast to the Telemark study, these studies have not included register data or advanced modelling of environmental exposure.

DETAILED DESCRIPTION:
Hypotheses and choice of methods:

Primary objective:

To identify preventive and health promoting measures for obstructive respiratory disease in a 5-year follow up of adults from the general population in Telemark.

Secondary objectives:

* Identify occupational risk factors for obstructive respiratory disease
* Assess interactions between risk factors and the individual
* Transfer relevant knowledge and advice regarding preventive and health promoting measures to individuals, health care professionals and authorities.

Research problems/questions (Q):

Q1 What are the emerging occupational risk factors for respiratory health? Q2 What are the social inequity/socioeconomic factors predicting respiratory disease? Q3 How does HRQoL develop over time? Q4 Do risk factors interact and how do they relate to the individual? Q5 What is the population attributable risk (PAR) for the identified risk factors, and what are the key factors for better prevention and respiratory health promotion?

Choice of methods/work packages (WP) and approaches (A):

WP I Occupational risk factors Q1 Emerging occupational causes and risk factors for respiratory disease and exacerbation

* A1.1 Assess associations between self-report of occupational exposure and new-onset and exacerbation of respiratory symptoms and diseases
* A1.2 Assess associations between job-exposure-matrix data (JEM) and new-onset and exacerbation of respiratory symptoms and diseases

WP II Individual risk factors Q2 Risk factors for social inequity in respiratory health

• A2.1 Assessment of the association between socio-demographic variables (gender, age, education, occupation and income) and respiratory health

WP III Complex interactions Q3 Health related quality of life development over time.

* A3.1 Impact of respiratory health and disease development and treatment on HRQoL development Q4 Interactions between risk factors and the individual
* A4.1 Identify interactions between risk factors and the individual by using advanced mathematical modelling Q5 The population attributable risk (PAR) for identified risk factors and key factors for better prevention and respiratory health promotion
* A5.1 Calculate PAR for risk factors identified in WP1-3 separately and combined
* A5.2 Based on PAR, estimate key factors for prevention and their cost

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma
* Controls without physician-diagnosed asthma

Exclusion Criteria:

* inability to fill-inn the questionnaire

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The researchers collected data in 2013 on respiratory symptoms and physician diagnosed asthma from 16.099 inhabitants of Telemark County (the cross-sectional baseline study called The Telemark-study I). A random sample from the baseline study of approximately 650 asthma cases and 650 controls were asked to take part in a medical examination in a case-control study in 2014-15.
  The five year follow up of the baseline (The Telemark-study II) study was performed in 2018 and included 13500 subjects. The follow-up of the nested case-control study started in September 2018 and is on-going.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurence of asthma and the association to specific occupational and environmental exposures and comorbidity | Five years
  Incidence and associations

SECONDARY OUTCOMES:
Risk factors for the occurence of asthma symptoms in subjects with asthma symptoms but no asthma diagnosis | Five years
  Odds ratio
Differences in lung function, FeNO and inflammatory markers in blood in asthma patients and the association of these changes to specific occupational and environmental exposures. | Five years
  Lung function indices, serum levels in blood

CONTACTS AND LOCATIONS:
Overall Officials: Johny Kongerud, Professor, Study Director — Oslo University, Oslo University Hospital; Anne Kristin Møller Fell, PhD, Principal Investigator — Sykehuset Telemark
Locations (1):
- Telemark Hospital, dep. of Occupational and Environmental Medicine, Skien, Telemark, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lillienberg L, Andersson E, Janson C, Dahlman-Hoglund A, Forsberg B, Holm M, Glslason T, Jogi R, Omenaas E, Schlunssen V, Sigsgaard T, Svanes C, Toren K. Occupational exposure and new-onset asthma in a population-based study in Northern Europe (RHINE). Ann Occup Hyg. 2013 May;57(4):482-92. doi: 10.1093/annhyg/mes083. Epub 2012 Dec 1. PMID 23204511
- [Background] de Vocht F, Zock JP, Kromhout H, Sunyer J, Anto JM, Burney P, Kogevinas M. Comparison of self-reported occupational exposure with a job exposure matrix in an international community-based study on asthma. Am J Ind Med. 2005 May;47(5):434-42. doi: 10.1002/ajim.20154. PMID 15828067
- [Background] Delclos GL, Gimeno D, Arif AA, Benavides FG, Zock JP. Occupational exposures and asthma in health-care workers: comparison of self-reports with a workplace-specific job exposure matrix. Am J Epidemiol. 2009 Mar 1;169(5):581-7. doi: 10.1093/aje/kwn387. Epub 2009 Jan 6. PMID 19126585
- [Derived] Fell AKM, Svendsen MV, Kim JL, Abrahamsen R, Henneberger PK, Toren K, Blanc PD, Kongerud J. Exposure to second-hand tobacco smoke and respiratory symptoms in non-smoking adults: cross-sectional data from the general population of Telemark, Norway. BMC Public Health. 2018 Jul 6;18(1):843. doi: 10.1186/s12889-018-5771-4. PMID 29980242